CLINICAL TRIAL: NCT04489303
Title: Virtual Patient Behavioral Response Training for Family Caregivers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Photozig, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Pz-A107a
Record Dates: First submitted 2020-07-24; First posted 2020-07-28 (Actual); Results first posted 2023-05-18 (Actual); Last update posted 2023-05-18 (Actual); Status verified 2023-05

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Patient Behavioral Response Training (Experimental): Caring Response mobile app with a behavioral training.
  Interventions: Behavioral: Caring Response App
- Educational Training (Active Comparator): Traditional educational program.
  Interventions: Behavioral: Traditional Educational/Resources Program

INTERVENTIONS:
Behavioral: Caring Response App — Participants will receive the Caring Response mobile app containing the Virtual Patient Behavioral Response Training.
  Arms: Virtual Patient Behavioral Response Training
Behavioral: Traditional Educational/Resources Program — Participants will receive a traditional educational/resources program, containing a workbook and online resources.
  Arms: Educational Training

SUMMARY:
Our study is designed to help caregivers of someone with Alzheimer's Disease and related dementia to understand and deal with the difficult behaviors of a person with dementia.

DETAILED DESCRIPTION:
The goal of this study is to develop and evaluate the Caring Response mobile app, containing a training that builds skills and stimulates practice. The investigators are evaluating different materials, which may encourage caregiver participation, enable user interaction, and promote better assimilation of concepts. The research team is designing the program to help to enhance caregivers' skills to deal with difficult behaviors, reduce distress, and improve quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Care for an individual with Alzheimer's Disease or other dementia.
* Own a smartphone or tablet and have Internet access.
* Minimum age of 18 years old.
* Spend at least 8 hours/week caring for a person with dementia.

Exclusion Criteria:

* Severe psychological or physical illness.
* Inability to read and follow English instructions.
* High level of depressive symptoms.
* Unwillingness to participate in all aspects of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2020-05-15 (Actual); Primary Completion 2021-05-30 (Actual); Study Completion 2021-05-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Kajiyama, MS, Principal Investigator — Photozig, Inc.
Locations (1):
- Photozig, Inc., Mountain View, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Virtual Patient Behavioral Response Training | Educational Training
Started | 78 | 78
Completed | 60 | 55
Not Completed | 18 | 23

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Virtual Patient Behavioral Response Training | Educational Training | Total
Number analyzed (Participants) | 78 | 78 | 156
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.0 (13.5) | 51.2 (14.1) | 48.6 (14.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60 | 64 | 124
  Male | 18 | 14 | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 14 | 18
  Not Hispanic or Latino | 74 | 64 | 138
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Revised Memory and Behavior Problems Checklist
Description: This scale measures the type/number of dementia patients disturbing behaviors, and how much they bother caregivers with 24 items describing possible troublesome behaviors that the patient might evidence in the past month. Caregivers are first asked whether the dementia patient had displayed any of these in the time period, and secondly to rate on a 5-point scale (0=not at all; 4= extremely) how much this "bothered or upset" them. A "conditional bother" score is calculated which is the "upset" or "bother" ratings for only the problematic behavior that occurred. The scale refers to the caregiver. Minimum score (best value)=0. Maximum score (worst value)=4. Higher values represent a worse outcome.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Virtual Patient Behavioral Response Training | Educational Training
Number analyzed (Participants) | 60 | 55
units on a scale | 0.66 (0.69) | 0.89 (0.78)

2. Primary Outcome: Center for Epidemiological Studies Depression Scale
Description: The Center for Epidemiological Studies Depression scale (CES-D) is a 20-item measure that asks about the frequency of depressive symptoms (affective, psychological, and somatic) within the past week.The scale refers to the caregiver. Minimum score (best value)=0. Maximum score (worst value)=60. Higher values represent a worse outcome.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Virtual Patient Behavioral Response Training | Educational Training
Number analyzed (Participants) | 60 | 55
units on a scale | 15.84 (9.97) | 21.00 (11.76)

3. Primary Outcome: Perceived Stress Scale
Description: The "Perceived Stress Scale" measures the overall level of stress. This instrument contains 10 items accessing overall appraisals of stress in the past month. The scale refers to the caregiver. Minimum score (best value)=0. Maximum score (worst value)=40. Higher values represent a worse outcome.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Virtual Patient Behavioral Response Training | Educational Training
Number analyzed (Participants) | 60 | 55
units on a scale | 15.78 (6.23) | 19.01 (7.09)

ADVERSE EVENTS:
Time Frame: 3 months
Description: The definitions are the same as the ones from clinicaltrials.gov
Arm/Group | Virtual Patient Behavioral Response Training | Educational Training
All-Cause Mortality (participants affected / at risk) | 0/78 | 0/78
Serious Adverse Events (participants affected / at risk) | 0/78 | 0/78
Other Adverse Events (participants affected / at risk) | 0/78 | 0/78

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-13): https://cdn.clinicaltrials.gov/large-docs/03/NCT04489303/Prot_SAP_000.pdf